CLINICAL TRIAL: NCT04230213
Title: A RANDOMIZED COMPARATIVE STUDY ASSESSING THE SWITCHING BETWEEN PF-06410293 AND HUMIRA (REGISTERED) IN COMBINATION WITH METHOTREXATE IN PARTICIPANTS WITH MODERATELY TO SEVERELY ACTIVE RHEUMATOID ARTHRITIS
Brief Title: A Comparative Study Between PF-06410293 and Humira® in Combination With Methotrexate in Participants With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B5381012; 2019-000284-24 (EudraCT Number); B5381012 (Other: Alias Study Number)
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Results first posted 2022-08-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — PF-06410293; Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm 1 (Experimental): Subcutaneous (SC) injection given every other week
  Interventions: Drug: PF-06410293; Drug: adalimumab
- Treatment Arm 2 (Active Comparator): SC injection given every other week
  Interventions: Drug: adalimumab

INTERVENTIONS:
Drug: PF-06410293 — SC injection
  Arms: Treatment Arm 1
Drug: adalimumab — SC injection
  Other Names: Humira ®

SUMMARY:
The study will assess the impact of pharmacokinetics (PK), safety and immunogenicity after switches between PF-06410293 and adalimumab and with continuous dosing with adalimumab in combination with methotrexate in subjects with moderately to severely active rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA based on 2010 ACR/EULAR for RA for at least a 4 month duration.
* Moderately to severely active RA based on local standard of care.

Exclusion Criteria:

-Evidence of untreated or inadequately treated latent or active TB.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (72):
- United States (4):
  - Graves Gilbert Clinic, Bowling Green, Kentucky
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Metroplex Clinical Research Center, Dallas, Texas
  - Rheumatology and Pulmonary Clinic, Beckley, West Virginia
- Bosnia and Herzegovina (4):
  - University Clinical Center of the Republic of Srpska, Banja Luka
  - Health Center Gradiska, Gradiška
  - Clinical Center University of Sarajevo, Sarajevo
  - General Hospital Prim. Dr.Abdulah Nakas, Sarajevo
- Bulgaria (3):
  - UMHAT "Dr Georgi Stranski" EAD, Pleven
  - DCC Sveti Georgi, Plovdiv
  - Unimed Medical Centre, Plovdiv
- Czechia (21):
  - IMEDICA s.r.o., Brno
  - Lekarna Na Lidicke, Brno
  - Lekarna Biovita, Brno
  - X-Medica, s.r.o., Brno
  - Revmacentrum MUDr. Mostera, s.r.o., Brno
  - L.K.N. Arthrocentrum, s.r.o., Hlučín
  - Plicni ambulance, Hlučín
  - Chirurgie Sibenik, Olomouc
  - CTCenter MaVe s.r.o, Olomouc
  - Lekarna u Pottingea, Olomouc
  - Lekarna Vesalion, Ostrava
  - CCR Czech a.s., Pardubice
  - Lekarna BENU, Pardubice
  - Lekarna Pod Platany, Prague
  - Revmatologicky ustav, Prague
  - CCR Prague s.r.o., Prague
  - Diagnostické centrum Olšanská s.r.o., Prague
  - Fakultni Nemocnice v Motole, Prague
  - Lekarna Hradebni s.r.o., Uherské Hradiště
  - MEDICAL PLUS s.r.o., Uherské Hradiště
  - Radiodiagnosticka ordinace a pracoviste, Uherské Hradiště
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences, Kauno klinikos, Kaunas
  - Klaipeda University Hospital, Klaipėda
- Poland (10):
  - Gabinet Internistyczno-Reumatologiczny Piotr Adrian Klimiuk, Bialystok
  - NZOZ Osteo-Medic s.c. A.Racewicz, J. Supronik, Bialystok
  - Małopolskie Badania Kliniczne Sp. z o. o. Sp. k., Krakow
  - Pratia MCM Krakow, Krakow
  - Zespol Poradni Specjalistycznych REUMED, Lublin
  - NZOZ Lecznica MAK-MED s.c., Nadarzyn
  - Twoja Przychodnia Centrum Medyczne Nowa Sol, Nowa Sól
  - Prywatna Praktyka Lekarska Prof. UM dr hab. med. Pawel Hrycaj, Poznan
  - Nasz Lekarz Przychodnie Medyczne, Torun
  - Rheuma Medicus Zaklad Opieki Zdrowotnej, Warsaw
- Russia (12):
  - Limited Liability Company "Clinic on Maroseyka", Moscow
  - Limited Liability Company Consultative and Diagnostic Rheumatological Center "Healthy Joints", Novosibirsk
  - FGBOU VO "Orenburg State Medical University" of the Ministry of Health of the Russian Federation, Orenburg
  - GBUZ "Orenburg Regional Clinical Hospital", Orenburg
  - SBHI of the Republic of Karelia "Republican Hospital n. a. V.A. Baranov", Petrozavodsk
  - FSBEI of HE "Ryazan State Medical University n. a academician I.P.Pavlov", Ryazan
  - SBI of the Ryazan Region "Regional Clinical Cardiology dispensary", Ryazan
  - SBI of Ryazan Region "Regional Clinical Hospital", Ryazan
  - Smolensk Regional Clinical Hospital, Smolensk
  - FSBEI of HE "Smolensk State Medical University" of the Ministry of Health of the RF, Smolensk
  - LLC "BioMed", Vladimir
  - LLC "Center for Medical Advice and Research-PRACTICE", Yaroslavl
- Serbia (3):
  - Institute of Rheumatology, Belgrade
  - Institute for Treatment and Rehabilitation Niska Banja, Niška Banja
  - Special Hospital for Rheumatic Diseases Novi Sad, Novi Sad
- South Africa (5):
  - Emmed Research, Pretoria, Gauteng
  - Jakaranda Hospital, Pretoria, Gauteng
  - Arthritis Clinical Research Trials, Cape Town, Western Cape
  - Panorama Medical Centre, Cape Town, Western Cape
  - Winelands Medical Research Centre, Stellenbosch, Western Cape
- Ukraine (8):
  - Komunalne nekomertsiine pidpryiemstvo Kharkivskoi oblasnoi rady Oblasna klinichna likarnia, Kharkiv
  - Medychnyi tsentr tovarystva z obmezhenoiu vidpovidalnistiu " Instytut revmatolohii ", Kyiv
  - Derzhavna ustanova Natsionalnyi naukovyi tsentr Instytut kardiolohii imeni akademika M.D. Strazheska, Kyiv
  - Komunalne Nekomertsiine Pidpryiemstvo "Tsentralna Miska Klinichna Likarnia, M. Ivano-Frankivsk
  - Komunalne nekomertsiine pidpryiemstvo "Odeska oblasna klinichna likarnia", Odesa
  - Bahatoprofilnyi medychnyi tsentr Odeskoho natsionalnoho medychnoho universytetu, Odesa
  - Komunalne nekomertsiine pidpryiemstvo "Vinnytska oblasna klinichna likarnia im. M.I. Pyrohova, Vinnytsia
  - Komunalne pidpryiemstvo "Likarnia No 1" Zhytomyrskoi miskoi rady, Zhytomyr

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Fleischmann RM, Saikali W, Lakhanpal S, Alvarez DF, Cox DS, Ianos CA, Zhang W, Cronenberger C, Wang K. Multiple switching between the biosimilar adalimumab PF-06410293 and reference adalimumab in patients with active rheumatoid arthritis: a phase 3, open-label, randomised, parallel-group study. Lancet Rheumatol. 2023 Sep;5(9):e532-e541. doi: 10.1016/S2665-9913(23)00161-3. Epub 2023 Aug 21. PMID 38251497
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B5381012

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 455 participants were enrolled in the study of which 10 participants were excluded from all the data analyses due to violation of Good Clinical Practice (GCP) principles. These 10 participants were not included in any section of results.
Groups:
- Humira (Adalimumab): All participants received Humira 40 milligrams (mg) once every 2 weeks subcutaneously for 10 weeks during Treatment Period 1 (TP1).
- Switching Arm: Humira and PF-06410293 (Adalimumab): Participants after completing TP1, were randomized to receive PF-06410293 40 mg once every 2 weeks subcutaneously for 6 weeks during Treatment Period 2 (TP2). TP2 was followed by Treatment Period 3 (TP3). In TP3 participants received Humira 40 mg once every 2 weeks subcutaneously for another 6 weeks. TP3 was followed by Treatment Period 4 (TP4). In TP4 participants received PF-06410293 40 mg once every 2 weeks subcutaneously for next 10 weeks. Participants were followed for 4 weeks post last dose.
- Non-switching Arm: Humira (Adalimumab): Participants after completing TP1, were randomized to continue treatment with Humira 40 mg once every 2 weeks subcutaneously for 22 weeks (during TP2 to TP4). Participants were followed for 4 weeks post last dose.
Period: TP1: Week 0 (Day 1) to Week 10
Arm/Group | Humira (Adalimumab) | Switching Arm: Humira and PF-06410293 (Adalimumab) | Non-switching Arm: Humira (Adalimumab)
Started | 445 | 0 | 0
Completed | 427 | 0 | 0
Not Completed | 18 | 0 | 0
Not completed — Other | 8 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 0 | 0
Not completed — Physician Decision | 3 | 0 | 0
Period: TP2: Week 10 to Week 16
Arm/Group | Humira (Adalimumab) | Switching Arm: Humira and PF-06410293 (Adalimumab) | Non-switching Arm: Humira (Adalimumab)
Started | 0 (TP1 ended when participants were randomized to Switching and Non-switching Arms) | 213 (Participants who completed TP1 were randomized to Switching arm.) | 214 (Participants who completed TP1 were randomized to Non-switching arm.)
Completed | 0 | 211 | 211
Not Completed | 0 | 2 | 3
Not completed — Other | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2
Period: TP3: Week 16 to Week 22
Arm/Group | Humira (Adalimumab) | Switching Arm: Humira and PF-06410293 (Adalimumab) | Non-switching Arm: Humira (Adalimumab)
Started | 0 | 211 | 211
Completed | 0 | 210 | 204
Not Completed | 0 | 1 | 7
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Other | 0 | 1 | 3
Period: TP4: Week 22 to Week 32
Arm/Group | Humira (Adalimumab) | Switching Arm: Humira and PF-06410293 (Adalimumab) | Non-switching Arm: Humira (Adalimumab)
Started | 0 | 210 | 204
Completed | 0 | 202 | 196
Not Completed | 0 | 8 | 8
Not completed — Other | 0 | 5 | 5
Not completed — Withdrawal by Subject | 0 | 1 | 2
Not completed — Physician Decision | 0 | 2 | 1
Period: Follow up: Week 32 to Week 36
Arm/Group | Humira (Adalimumab) | Switching Arm: Humira and PF-06410293 (Adalimumab) | Non-switching Arm: Humira (Adalimumab)
Started | 0 | 202 | 196
Completed | 0 | 201 | 194
Not Completed | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Other | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all the participants who were enrolled in TP1.
Groups:
- Humira (Adalimumab): All participants received Humira 40 mg once every 2 weeks subcutaneously for 10 weeks during TP1. After completing TP1, participants were randomized to Switching Arm: Humira and PF-06410293 (Adalimumab) and Non-switching Arm: Humira (Adalimumab). Participants randomized to Switching Arm: Humira and PF-06410293 (Adalimumab) received PF-06410293 40 mg once every 2 weeks subcutaneously for 6 weeks during TP2. TP2 was followed by TP3. In TP3 participants received Humira 40 mg once every 2 weeks subcutaneously for another 6 weeks. TP3 was followed by TP4. In TP4 participants received PF-06410293 40 mg once every 2 weeks subcutaneously for next 10 weeks. Participants randomized to Non-switching Arm: Humira (Adalimumab) after completing TP1 continued treatment with Humira 40 mg once every 2 weeks subcutaneously for 22 weeks (during TP2 to TP4). Participants were followed for 4 weeks post last dose.
Arm/Group | Humira (Adalimumab)
Number analyzed (Participants) | 445
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Here, number analyzed signifies number of participants evaluable for specified rows i.e. Humira (adalimumab) arm including all participants enrolled in TP1 and Switching arm: Humira and PF-06410293 (Adalimumab) and Non-switching Arm: Humira (Adalimumab) arms including all participants who were randomized at Week 10.
  Years
    Lead-In TP1: Humira (Adalimumab) | 53.60 (11.17)
    Switching arm: Humira and PF-06410293 (Adalimumab): number analyzed (Participants) | 213
    Switching arm: Humira and PF-06410293 (Adalimumab) | 53.60 (11.26)
    Non-Switching arm: Humira (Adalimumab): number analyzed (Participants) | 214
    Non-Switching arm: Humira (Adalimumab) | 53.35 (11.30)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Here, number analyzed signifies number of participants evaluable for specified rows i.e. Humira (adalimumab) arm including all participants enrolled in TP1 and Switching arm: Humira and PF-06410293 (Adalimumab) and Non-switching Arm: Humira (Adalimumab) arms including all participants who were randomized at Week 10.
  Participants
    Lead-In TP1: Humira (Adalimumab): Female | 368
    Lead-In TP1: Humira (Adalimumab): Male | 77
    Switching arm: Humira and PF-06410293 (Adalimumab): number analyzed (Participants) | 213
    Switching arm: Humira and PF-06410293 (Adalimumab): Female | 175
    Switching arm: Humira and PF-06410293 (Adalimumab): Male | 38
    Non-Switching arm: Humira (Adalimumab): number analyzed (Participants) | 214
    Non-Switching arm: Humira (Adalimumab): Female | 179
    Non-Switching arm: Humira (Adalimumab): Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Here, number analyzed signifies number of participants evaluable for specified rows i.e. Humira (adalimumab) arm including all participants enrolled in TP1 and Switching arm: Humira and PF-06410293 (Adalimumab) and Non-switching Arm: Humira (Adalimumab) arms including all participants who were randomized at Week 10.
  Participants
    Lead-In TP1: Humira (Adalimumab): Hispanic or Latino | 4
    Lead-In TP1: Humira (Adalimumab): Not Hispanic or Latino | 440
    Lead-In TP1: Humira (Adalimumab): Unknown or Not Reported | 1
    Switching arm: Humira and PF-06410293 (Adalimumab): number analyzed (Participants) | 213
    Switching arm: Humira and PF-06410293 (Adalimumab): Hispanic or Latino | 2
    Switching arm: Humira and PF-06410293 (Adalimumab): Not Hispanic or Latino | 210
    Switching arm: Humira and PF-06410293 (Adalimumab): Unknown or Not Reported | 1
    Non-Switching arm: Humira (Adalimumab): number analyzed (Participants) | 214
    Non-Switching arm: Humira (Adalimumab): Hispanic or Latino | 1
    Non-Switching arm: Humira (Adalimumab): Not Hispanic or Latino | 213
    Non-Switching arm: Humira (Adalimumab): Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Here, number analyzed signifies number of participants evaluable for specified rows i.e. Humira (adalimumab) arm including all participants enrolled in TP1 and Switching arm: Humira and PF-06410293 (Adalimumab) and Non-switching Arm: Humira (Adalimumab) arms including all participants who were randomized at Week 10.
  Participants
    Lead-In TP1: Humira (Adalimumab): American Indian or Alaska Native | 0
    Lead-In TP1: Humira (Adalimumab): Asian | 0
    Lead-In TP1: Humira (Adalimumab): Native Hawaiian or Other Pacific Islander | 0
    Lead-In TP1: Humira (Adalimumab): Black or African American | 2
    Lead-In TP1: Humira (Adalimumab): White | 440
    Lead-In TP1: Humira (Adalimumab): More than one race | 0
    Lead-In TP1: Humira (Adalimumab): Unknown or Not Reported | 3
    Switching arm: Humira and PF-06410293 (Adalimumab): number analyzed (Participants) | 213
    Switching arm: Humira and PF-06410293 (Adalimumab): American Indian or Alaska Native | 0
    Switching arm: Humira and PF-06410293 (Adalimumab): Asian | 0
    Switching arm: Humira and PF-06410293 (Adalimumab): Native Hawaiian or Other Pacific Islander | 0
    Switching arm: Humira and PF-06410293 (Adalimumab): Black or African American | 0
    Switching arm: Humira and PF-06410293 (Adalimumab): White | 212
    Switching arm: Humira and PF-06410293 (Adalimumab): More than one race | 0
    Switching arm: Humira and PF-06410293 (Adalimumab): Unknown or Not Reported | 1
    Non-Switching arm: Humira (Adalimumab): number analyzed (Participants) | 214
    Non-Switching arm: Humira (Adalimumab): American Indian or Alaska Native | 0
    Non-Switching arm: Humira (Adalimumab): Asian | 0
    Non-Switching arm: Humira (Adalimumab): Native Hawaiian or Other Pacific Islander | 0
    Non-Switching arm: Humira (Adalimumab): Black or African American | 0
    Non-Switching arm: Humira (Adalimumab): White | 210
    Non-Switching arm: Humira (Adalimumab): More than one race | 2
    Non-Switching arm: Humira (Adalimumab): Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Serum Concentration (Cmax) of Adalimumab
Description: Cmax refers to maximum observed serum concentration of drug. The geometric coefficient of variation is expressed in percentage.
Time Frame: Pre-dose, 48, 72, 96, 144, 240 and 336 hours post dose on Day 211 (Week 30)
Population: Pharmacokinetic (PK) population included all randomized participants who were dosed to initiate the week 30 steady-state PK profile and remained on background methotrexate with no major protocol deviations influencing the PK assessment. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. Since time points for analysis for this outcome measure were falling in TP4, hence only switching and non-switching arms data were reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Switching Arm: Humira and PF-06410293 (Adalimumab) | Non-switching Arm: Humira (Adalimumab)
Number analyzed (Participants) | 194 | 186
Micrograms per milliliter | 9.156 (97) | 8.974 (97)
Statistical Analysis 1: Comparison: Switching Arm: Humira and PF-06410293 (Adalimumab) vs Non-switching Arm: Humira (Adalimumab); Test type: Equivalence — Equivalence was to be determined if the 90% confidence interval of the geometric mean ratio falls within the 80% to 125% range; Geometric mean ratio (percentage) = 102.56, 90% CI 2-sided [89.78 to 117.17] — Analysis was performed using analysis of variance (ANOVA) model

2. Primary Outcome: Area Under the Serum Concentration-Time Curve Over the Dosing Interval (AUCtau) of Adalimumab
Description: Area under the serum concentration curve from time 0 to end of dosing interval (tau), where dosing interval was once every two weeks. The geometric coefficient of variation is expressed in percentage.
Time Frame: Pre-dose, 48, 72, 96, 144, 240 and 336 hours post dose on Day 211 (Week 30)
Population: PK population included all randomized participants who were dosed to initiate the Week 30 steady-state PK profile and remained on background methotrexate with no major protocol deviations influencing the PK assessment. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. Since time points for analysis for this outcome measure were falling in TP4, hence only switching and non-switching arms data were reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms*hour per milliliter
Arm/Group | Switching Arm: Humira and PF-06410293 (Adalimumab) | Non-switching Arm: Humira (Adalimumab)
Number analyzed (Participants) | 189 | 183
Micrograms*hour per milliliter | 2472 (129) | 2365 (133)
Statistical Analysis 1: Comparison: Switching Arm: Humira and PF-06410293 (Adalimumab) vs Non-switching Arm: Humira (Adalimumab); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric mean ratio (Percentage) = 105.31, 90% CI 2-sided [89.16 to 124.39] — Analysis was performed using ANOVA model

3. Secondary Outcome: Time to Reach Cmax (Tmax) of Adalimumab
Description: Tmax is the time taken (in hours) to reach the maximum serum drug concentration.
Time Frame: Pre-dose, 48, 72, 96, 144, 240 and 336 hours post dose on Day 211 (Week 30)
Population: PK population included all randomized participants who were dosed to initiate the Week 30 steady state PK profile and remained on background methotrexate with no major protocol deviations influencing the PK assessment. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. Since time points for analysis for this outcome measure were falling in TP4, hence only switching and non-switching arms data were reported.
Measure: Median (Full Range); unit: Hours
Arm/Group | Switching Arm: Humira and PF-06410293 (Adalimumab) | Non-switching Arm: Humira (Adalimumab)
Number analyzed (Participants) | 194 | 186
Hours | 71.80 [0.000 to 336] | 72.00 [0.000 to 337]

4. Secondary Outcome: Average Serum Concentration (Cav) of Adalimumab
Description: Cav was defined as average serum concentration over the dosing interval. The geometric coefficient of variation is expressed in percentage.
Time Frame: Pre-dose, 48, 72, 96, 144, 240 and 336 hours post dose on Day 211 (Week 30)
Population: PK population included all randomized participants who were dosed to initiate the Week 30 steady state PK profile and remained on background methotrexate with no major protocol deviations influencing the PK assessment. Here 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure. Since time points for analysis for this outcome measure were falling in TP4, hence only switching and non-switching arms data were reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Switching Arm: Humira and PF-06410293 (Adalimumab) | Non-switching Arm: Humira (Adalimumab)
Number analyzed (Participants) | 189 | 183
Micrograms per milliliter | 7.357 (130) | 7.040 (133)

5. Secondary Outcome: Apparent Clearance (CL/F) of Serum Adalimumab
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. CL/F was calculated as dose administered divided by area under the concentration curve from time 0 extrapolated to infinite time (AUCinf). The geometric coefficient of variation is expressed in percentage.
Time Frame: Pre-dose, 48, 72, 96, 144, 240 and 336 hours post dose on Day 211 (Week 30)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliter per hour
Arm/Group | Switching Arm: Humira and PF-06410293 (Adalimumab) | Non-switching Arm: Humira (Adalimumab)
Number analyzed (Participants) | 189 | 183
Milliliter per hour | 16.19 (129) | 16.91 (133)

6. Secondary Outcome: Pre-dose Serum Concentration During Multiple Dosing (Ctrough) of Adalimumab
Description: Ctrough was defined as pre-dose serum concentration during multiple dosing and observed directly from data.
Time Frame: Pre-dose on Day 1, 71,113, 155, 169, 183, 197 and 211
Population: Safety randomized population included all participants who were randomized and received at least one dose of study treatment following the randomization at Study Week 10. Data for Days 1 and 71 were identified retrospectively for participants in the safety randomized population, hence included in the switching and non-switching reporting groups. Here, "Number Analyzed" signifies participants evaluable for each specified category.
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | Switching Arm: Humira and PF-06410293 (Adalimumab) | Non-switching Arm: Humira (Adalimumab)
Number analyzed (Participants) | 213 | 214
Micrograms per milliliter
  Day 1 | 0.03102 (0.15291) | 0.05703 (0.29719)
  Day 71: number analyzed (Participants) | 211 | 214
  Day 71 | 6.999 (4.4196) | 6.675 (4.3310)
  Day 113: number analyzed (Participants) | 210 | 209
  Day 113 | 7.763 (5.0812) | 7.374 (4.8807)
  Day 155: number analyzed (Participants) | 208 | 200
  Day 155 | 7.900 (5.2493) | 7.558 (5.0502)
  Day 169: number analyzed (Participants) | 204 | 197
  Day 169 | 7.918 (5.1756) | 7.767 (5.1860)
  Day 183: number analyzed (Participants) | 202 | 197
  Day 183 | 8.259 (5.3404) | 7.933 (5.1299)
  Day 197: number analyzed (Participants) | 204 | 197
  Day 197 | 8.347 (5.5458) | 8.022 (5.2046)
  Day 211: number analyzed (Participants) | 206 | 198
  Day 211 | 8.477 (5.4604) | 7.891 (5.1818)

7. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs and Treatment Related TEAEs: TP1
Description: An adverse event (AE) was any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An SAE was any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent or significant disability/ incapacity; congenital anomaly/birth defect and other important medical events. Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. TEAE for TP1 was defined as any AE that occurred after the beginning of study treatment in TP1 and before the first dose of study treatment administration after randomization in TP2. AEs included both serious and all non-serious AEs.
Time Frame: Day 1 up to maximum of 10 Weeks
Population: Safety population for TP1 included all participants who were enrolled and received at least one dose of study treatment in TP1.
Measure: Count of Participants; unit: Participants
Groups:
- Humira (Adalimumab): All participants received Humira 40 mg once every 2 weeks subcutaneously for 10 weeks during TP1.
Arm/Group | Humira (Adalimumab)
Number analyzed (Participants) | 445
Participants
  TEAEs | 107
  Serious TEAEs | 13
  Treatment related TEAEs | 31

8. Secondary Outcome: Number of Participants With TEAEs, Serious TEAEs and Treatment Related TEAEs: TP2 and Beyond
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An SAE was any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent or significant disability/ incapacity; congenital anomaly/birth defect and other important medical events. Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. TEAE for TP2 and beyond was defined as any AE that occurred after administering the first dose of study treatment after randomization in TP2 and up to 4 weeks after last dose. AEs included both serious and all non-serious AEs.
Time Frame: Post randomization up to maximum of 4 weeks after last dose (maximum of 26 weeks)
Population: Safety randomized population included all participants who were randomized and received at least one dose of study treatment following the randomization at Study Week 10.
Measure: Count of Participants; unit: Participants
Arm/Group | Switching Arm: Humira and PF-06410293 (Adalimumab) | Non-switching Arm: Humira (Adalimumab)
Number analyzed (Participants) | 213 | 214
Participants
  TEAEs | 82 | 62
  Serious TEAEs | 3 | 8
  Treatment related TEAEs | 19 | 10

9. Secondary Outcome: Number of Participants With Grade 3 or Higher TEAEs: TP1
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. TEAE for TP1 was defined as any AE that occurred after the beginning of study treatment in TP1 and before the first dose of study treatment administration after randomization in TP2. AEs were graded using the Common Terminology Criteria for Adverse Events where, grade 1=mild AE; grade 2=moderate AE; grade 3=severe AE; grade 4= life-threatening consequences; urgent intervention indicated; and grade 5= death related to AE. Number of participants with grade 3 or higher TEAEs were presented.
Time Frame: Day 1 up to maximum of 10 Weeks
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Humira (Adalimumab)
Number analyzed (Participants) | 445
Participants | 14

10. Secondary Outcome: Number of Participants With Grade 3 or Higher TEAEs: TP2 and Beyond
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. TEAE for TP2 and beyond was defined as any AE that occurred after the first dose of study treatment administration after randomization in TP2 and up to 4 weeks after last dose. AEs were graded using the Common Terminology Criteria for Adverse Events where, grade 1=mild AE; grade 2=moderate AE; grade 3=severe AE; grade 4= life-threatening consequences; urgent intervention indicated; and grade 5= death related to AE. Number of participants with grade 3 or higher TEAEs were presented.
Time Frame: Post randomization up to maximum of 4 weeks after last dose (maximum of 26 weeks)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Switching Arm: Humira and PF-06410293 (Adalimumab) | Non-switching Arm: Humira (Adalimumab)
Number analyzed (Participants) | 213 | 214
Participants | 5 | 8

11. Secondary Outcome: Number of Participants Who Discontinued Treatment and Study Due to TEAEs: TP1
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. TEAE for TP1 was defined as any AE that occurred after the beginning of study treatment in TP1 and before the first dose of study treatment administration after randomization in TP2. Participants who discontinued treatment due to TEAEs were those who had an AE record indicating that action taken with study treatment was drug withdrawn but AE did not cause the participant to be discontinued from study. Participants who discontinued from study due to TEAE were those who had an TEAE in TP1 indicating that the AE caused the participant to be discontinued from the study.
Time Frame: Day 1 up to maximum of 10 Weeks
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Humira (Adalimumab)
Number analyzed (Participants) | 445
Participants
  Discontinued from treatment due to TEAEs | 3
  Discontinued from study due to TEAE | 12

12. Secondary Outcome: Number of Participants Who Discontinued Treatment and Study Due to TEAEs: TP2 and Beyond
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. TEAE for TP2 and beyond was defined as any AE that occurred after the first dose of study treatment administration after randomization in TP2 and up to 4 weeks after last dose. AEs included both serious and all non-serious AEs. Participants who discontinued treatment due to TEAEs were those who had an AE record indicating that action taken with study treatment was drug withdrawn but AE did not cause the participant to be discontinued from study. Participants who discontinued from study due to TEAE were those who had an AE record indicating that the AE caused the participant to be discontinued from the study.
Time Frame: Post randomization up to maximum of 4 weeks after last dose (maximum of 26 weeks)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Switching Arm: Humira and PF-06410293 (Adalimumab) | Non-switching Arm: Humira (Adalimumab)
Number analyzed (Participants) | 213 | 214
Participants
  Discontinued from treatment due to TEAEs | 0 | 3
  Discontinued from study due to TEAEs | 8 | 9

13. Secondary Outcome: Number of Participants With TEAEs of Special Interest: TP2 and Beyond
Description: AEs of special interest (AESI) included: hypersensitivity events (anaphylactic reaction, hypersensitivity, angioedema, delayed immune responses and injection site reactions [ISRs]); blood and lymphatic system events (white blood cell disorders and anemias nonhemolytic and marrow depression); cardiovascular events (cardiac failure, hypertension and myocardial infarction); demyelinating conditions, gastric/hepatic events (gastrointestinal perforation, ulceration, hemorrhage or obstruction and hepatic disorders); infections and infestations (including TB and other opportunistic infections); malignancies (neoplasms benign, malignant and unspecified [including cysts and polyps]) and lupus like syndrome. TEAE was defined as any AE that occurred after the first dose of study treatment administered after randomization in TP2. Number of participants with any AESI were presented in this outcome measure.
Time Frame: Post randomization up to maximum of 4 weeks after last dose (maximum of 26 weeks)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Switching Arm: Humira and PF-06410293 (Adalimumab) | Non-switching Arm: Humira (Adalimumab)
Number analyzed (Participants) | 213 | 214
Participants | 58 | 47

14. Secondary Outcome: Number of Participants With Potential Immunogenic AEs to Study Treatment: TP2 and Beyond Among Anti-drug Antibody (ADA) Positive Participants During TP1
Description: In this outcome, participants who were antidrug antibody (ADA) positive during TP1 were assessed in TP2 and beyond per visit for their ADA status at the time of start of their potential immunogenic AEs including ISRs, medically evaluated board standard MedDRA query (SMQ) of potential hypersensitivity (anaphylactic reactions, hypersensitivity and angioedema), medically evaluated AEs meeting Sampson criteria, cytokine storm and delayed immune responses (DIR). ADA positive was defined as ADA titer >=1.88.
Time Frame: TP2 and Beyond: Week 16, 22, 24, 26, 28, 30, 32
Population: Safety randomized population included all participants who were randomized and received at least one dose of investigational product following the randomization at Study Week 10.Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. Here, "Number Analyzed" signifies participants evaluable for specific rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Switching Arm: Humira and PF-06410293 (Adalimumab) | Non-switching Arm: Humira (Adalimumab)
Number analyzed (Participants) | 55 | 59
Participants
  Week 16: ISR: number analyzed (Participants) | 55 | 57
  Week 16: ISR | 0 | 1
  Week 16: Medically evaluated Sampson criteria met: number analyzed (Participants) | 55 | 57
  Week 16: Medically evaluated Sampson criteria met | 0 | 0
  Week 16: AEs belonging to SMQ Group: number analyzed (Participants) | 55 | 57
  Week 16: AEs belonging to SMQ Group | 0 | 0
  Week 22: ISR: number analyzed (Participants) | 55 | 55
  Week 22: ISR | 0 | 1
  Week 22: Medically evaluated Sampson criteria met: number analyzed (Participants) | 55 | 55
  Week 22: Medically evaluated Sampson criteria met | 0 | 0
  Week 22: AEs belonging to SMQ Group: number analyzed (Participants) | 55 | 55
  Week 22: AEs belonging to SMQ Group | 0 | 0
  Week 24: ISR: number analyzed (Participants) | 55 | 54
  Week 24: ISR | 0 | 1
  Week 24: Medically evaluated Sampson criteria met: number analyzed (Participants) | 55 | 54
  Week 24: Medically evaluated Sampson criteria met | 0 | 0
  Week 24: AEs belonging to SMQ Group: number analyzed (Participants) | 55 | 54
  Week 24: AEs belonging to SMQ Group | 0 | 1
  Week 26: ISR: number analyzed (Participants) | 54 | 53
  Week 26: ISR | 1 | 1
  Week 26: Medically evaluated Sampson criteria met: number analyzed (Participants) | 54 | 53
  Week 26: Medically evaluated Sampson criteria met | 0 | 0
  Week 26: AEs belonging to SMQ Group: number analyzed (Participants) | 54 | 53
  Week 26: AEs belonging to SMQ Group | 0 | 0
  Week 28: ISR: number analyzed (Participants) | 55 | 53
  Week 28: ISR | 0 | 1
  Week 28: Medically evaluated Sampson criteria met: number analyzed (Participants) | 55 | 53
  Week 28: Medically evaluated Sampson criteria met | 0 | 0
  Week 28: AEs belonging to SMQ Group: number analyzed (Participants) | 55 | 53
  Week 28: AEs belonging to SMQ Group | 0 | 0
  Week 30: ISR: number analyzed (Participants) | 55 | 54
  Week 30: ISR | 0 | 1
  Week 30: Medically evaluated Sampson criteria met: number analyzed (Participants) | 55 | 54
  Week 30: Medically evaluated Sampson criteria met | 0 | 0
  Week 30: AEs belonging to SMQ Group: number analyzed (Participants) | 55 | 54
  Week 30: AEs belonging to SMQ Group | 1 | 0
  Week 32: ISR: number analyzed (Participants) | 54 | 59
  Week 32: ISR | 0 | 0
  Week 32: Medically evaluated Sampson criteria met: number analyzed (Participants) | 54 | 59
  Week 32: Medically evaluated Sampson criteria met | 0 | 0
  Week 32: AEs belonging to SMQ Group: number analyzed (Participants) | 54 | 59
  Week 32: AEs belonging to SMQ Group | 0 | 0

15. Secondary Outcome: Number of Participants With Potential Immunogenic AEs to Study Treatment: TP2 and Beyond Among ADA Negative Participants During TP1
Description: In this outcome, participants who were ADA negative during TP1 were assessed in TP2 and beyond per visit for their ADA status at the time of start of their potential immunogenic AEs including ISRs, medically evaluated board SMQ of potential hypersensitivity (anaphylactic reactions, hypersensitivity and angioedema), medically evaluated AEs meeting Sampson criteria, cytokine storm and DIR. ADA negative was defined as ADA titer <1.88.
Time Frame: TP2 and Beyond: Week 16, 22, 24, 26, 28, 30, 32
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Switching Arm: Humira and PF-06410293 (Adalimumab) | Non-switching Arm: Humira (Adalimumab)
Number analyzed (Participants) | 156 | 155
Participants
  Week 16: ISR: number analyzed (Participants) | 153 | 152
  Week 16: ISR | 4 | 2
  Week 16: Medically evaluated Sampson criteria met: number analyzed (Participants) | 153 | 152
  Week 16: Medically evaluated Sampson criteria met | 0 | 0
  Week 16: AEs belonging to SMQ Group: number analyzed (Participants) | 153 | 152
  Week 16: AEs belonging to SMQ Group | 0 | 0
  Week 22: ISR: number analyzed (Participants) | 151 | 147
  Week 22: ISR | 1 | 1
  Week 22: Medically evaluated Sampson criteria met: number analyzed (Participants) | 151 | 147
  Week 22: Medically evaluated Sampson criteria met | 0 | 0
  Week 22: AEs belonging to SMQ Group: number analyzed (Participants) | 151 | 147
  Week 22: AEs belonging to SMQ Group | 0 | 0
  Week 24: ISR: number analyzed (Participants) | 150 | 145
  Week 24: ISR | 0 | 2
  Week 24: Medically evaluated Sampson criteria met: number analyzed (Participants) | 150 | 145
  Week 24: Medically evaluated Sampson criteria met | 0 | 0
  Week 24: AEs belonging to SMQ Group: number analyzed (Participants) | 150 | 145
  Week 24: AEs belonging to SMQ Group | 0 | 0
  Week 26: ISR: number analyzed (Participants) | 148 | 145
  Week 26: ISR | 0 | 2
  Week 26: Medically evaluated Sampson criteria met: number analyzed (Participants) | 148 | 145
  Week 26: Medically evaluated Sampson criteria met | 0 | 0
  Week 26: AEs belonging to SMQ Group: number analyzed (Participants) | 148 | 145
  Week 26: AEs belonging to SMQ Group | 0 | 0
  Week 28: ISR: number analyzed (Participants) | 148 | 144
  Week 28: ISR | 0 | 1
  Week 28: Medically evaluated Sampson criteria met: number analyzed (Participants) | 148 | 144
  Week 28: Medically evaluated Sampson criteria met | 0 | 0
  Week 28: AEs belonging to SMQ Group: number analyzed (Participants) | 148 | 144
  Week 28: AEs belonging to SMQ Group | 0 | 0
  Week 30: ISR: number analyzed (Participants) | 149 | 144
  Week 30: ISR | 0 | 1
  Week 30: Medically evaluated Sampson criteria met: number analyzed (Participants) | 149 | 144
  Week 30: Medically evaluated Sampson criteria met | 0 | 0
  Week 30: AEs belonging to SMQ Group: number analyzed (Participants) | 149 | 144
  Week 30: AEs belonging to SMQ Group | 0 | 0
  Week 32: ISR: number analyzed (Participants) | 152 | 149
  Week 32: ISR | 0 | 1
  Week 32: Medically evaluated Sampson criteria met: number analyzed (Participants) | 152 | 149
  Week 32: Medically evaluated Sampson criteria met | 0 | 0
  Week 32: AEs belonging to SMQ Group: number analyzed (Participants) | 152 | 149
  Week 32: AEs belonging to SMQ Group | 0 | 0

16. Secondary Outcome: Number of Participants With TEAEs and Serious TEAEs Related to COVID-19: TP1
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An SAE was any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent or significant disability/ incapacity; congenital anomaly/birth defect and other important medical events. TEAE for TP1 was defined as any AE that occurred after the beginning of study treatment in TP1 and before the first dose of study treatment administration after randomization in TP2. AEs included both serious and all non-serious AEs. TEAEs and serious TEAEs related to Covid-19 as per investigator's assessment were presented.
Time Frame: Day 1 up to maximum of 10 Weeks
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Humira (Adalimumab)
Number analyzed (Participants) | 445
Participants
  TEAE | 10
  Serious TEAE | 6

17. Secondary Outcome: Number of Participants With TEAEs and Serious TEAEs Related to COVID-19: TP2 and Beyond
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An SAE was any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent or significant disability/ incapacity; congenital anomaly/birth defect and other important medical events. TEAE for TP2 and beyond was defined as any AE that occurred after the first dose of study treatment administration after randomization in TP2 and up to 4 weeks after last dose. AEs included both serious and all non-serious AEs. TEAEs and serious TEAEs related to Covid-19 as per investigator's assessment were presented.
Time Frame: Post randomization up to maximum of 4 weeks after last dose (maximum of 26 weeks)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Switching Arm: Humira and PF-06410293 (Adalimumab) | Non-switching Arm: Humira (Adalimumab)
Number analyzed (Participants) | 213 | 214
Participants
  TEAE | 20 | 16
  Serious TEAE | 1 | 3

18. Secondary Outcome: Number of Participants Who Discontinued Treatment and Study Due to TEAEs Related to COVID-19: TP1
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. TEAE for TP1 was defined as any AE that occurred after the beginning of study treatment in TP1 and before the first dose of study treatment administration after randomization in TP2. Participants who discontinued treatment due to TEAEs were those who had an AE record indicating that action taken with study treatment was drug withdrawn but AE did not cause the participant to be discontinued from study. Participants who discontinued from study due to TEAE were those who had an AE record indicating that the AE caused the participant to be discontinued from the study. TEAEs were related to Covid-19.
Time Frame: Day 1 up to maximum of 10 Weeks
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Humira (Adalimumab)
Number analyzed (Participants) | 445
Participants
  Discontinued from treatment due to TEAEs | 0
  Discontinued from study due to TEAE | 6

19. Secondary Outcome: Number of Participants Who Discontinued Treatment and Study Due to TEAEs Related to COVID-19: TP2 and Beyond
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. TEAE for TP2 and beyond was defined as any AE that occurred after the first dose of study treatment administration after randomization in TP2 and up to 4 weeks after last dose. AEs included both serious and all non-serious AEs. Participants who discontinued treatment due to TEAEs were those who had an AE record indicating that action taken with study treatment was drug withdrawn but AE did not cause the participant to be discontinued from study. Participants who discontinued from study due to TEAE were those who had an AE record indicating that the AE caused the participant to be discontinued from the study. TEAEs were related to Covid-19.
Time Frame: Post randomization up to maximum of 4 weeks after last dose (maximum of 26 weeks)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Switching Arm: Humira and PF-06410293 (Adalimumab) | Non-switching Arm: Humira (Adalimumab)
Number analyzed (Participants) | 213 | 214
Participants
  Discontinued from treatment due to TEAEs | 0 | 0
  Discontinued from study due to TEAE | 3 | 4

20. Secondary Outcome: Number of Participants With Laboratory Abnormalities: TP1
Description: Blood samples were collected for the analysis of following laboratory parameters: hematology parameters (hemoglobin, erythrocyte mean corpuscular volume, erythrocyte mean corpuscular hemoglobin, erythrocyte mean corpuscular hemoglobin concentration platelet count, leukocytes, lymphocytes, neutrophils, eosinophils, monocytes); clinical chemistry parameters (bilirubin, alanine aminotransferase [ALT], blood urea nitrogen [BUN], creatinine, potassium, bicarbonate); urine parameters: urine protein, urine hemoglobin, nitrite, leukocyte esterase and bacteria. Number of participants with any laboratory abnormalities is presented.
Time Frame: Day 1 up to maximum of 10 Weeks
Population: Safety population for TP1 included all participants who were enrolled and received at least one dose of study treatment in TP1. Here 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Humira (Adalimumab)
Number analyzed (Participants) | 437
Participants | 134

21. Secondary Outcome: Number of Participants With Laboratory Abnormalities: TP2 and Beyond
Description: Blood samples were collected for the analysis of following laboratory parameters: hematology parameters (hemoglobin, erythrocyte mean corpuscular volume, erythrocyte mean corpuscular hemoglobin, erythrocyte mean corpuscular hemoglobin concentration platelet count, leukocytes, lymphocytes, neutrophils, eosinophils, monocytes); clinical chemistry parameters (bilirubin, ALT, BUN, creatinine, potassium, bicarbonate); urine parameters: urine protein, urine hemoglobin, nitrite, leukocyte esterase and bacteria. Number of participants with any laboratory abnormalities is presented.
Time Frame: Post randomization up to end of study treatment (maximum of 22 weeks)
Population: Safety randomized population included all participants who were randomized and received at least one dose of dose of investigational product following the randomization at Study Week 10. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Switching Arm: Humira and PF-06410293 (Adalimumab) | Non-switching Arm: Humira (Adalimumab)
Number analyzed (Participants) | 211 | 208
Participants | 71 | 83

22. Secondary Outcome: Number of Participants With Hematology Results by Maximum Common Toxicity Criteria (CTC) Grade: TP2 and Beyond
Description: Blood samples were collected for the analysis of following hematology parameters: anemia, hemoglobin increased, leukocytosis, lymphocyte count decreased, lymphocyte count increased, neutrophil count decreased, platelet count decreased, white blood cell decreased. Laboratory parameters were graded according to National Cancer Institute-CTC version 4.03 where, Grade 0= within normal limits; Grade1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences and Grade 5: death. Categories with at least 1 non-zero value were reported in this outcome measure.
Time Frame: Post randomization up to end of study treatment (maximum of 22 weeks)
Population: Safety randomized population included all participants who were randomized and received at least one dose of dose of investigational product following the randomization at Study Week 10. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. Here, "Number Analyzed" signifies participants evaluable for each row.
Measure: Count of Participants; unit: Participants
Arm/Group | Switching Arm: Humira and PF-06410293 (Adalimumab) | Non-switching Arm: Humira (Adalimumab)
Number analyzed (Participants) | 209 | 205
Participants
  Grade 0: Anemia | 198 | 190
  Grade 0: Hemoglobin increased | 207 | 201
  Grade 0: Leukocytosis | 209 | 205
  Grade 0: Lymphocyte count decreased | 204 | 200
  Grade 0: Lymphocyte count increased | 203 | 196
  Grade 0: Neutrophil count decreased: number analyzed (Participants) | 209 | 204
  Grade 0: Neutrophil count decreased | 198 | 197
  Grade 0: Platelet count decreased: number analyzed (Participants) | 207 | 204
  Grade 0: Platelet count decreased | 201 | 200
  Grade 0: White blood cell decreased | 202 | 199
  Grade 1: Anemia | 5 | 7
  Grade 1: Hemoglobin increased | 2 | 3
  Grade 1: Lymphocyte count decreased | 4 | 3
  Grade 1: Neutrophil count decreased: number analyzed (Participants) | 209 | 204
  Grade 1: Neutrophil count decreased | 4 | 3
  Grade 1: Platelet count decreased: number analyzed (Participants) | 207 | 204
  Grade 1: Platelet count decreased | 6 | 4
  Grade 1: White blood cell decreased | 6 | 6
  Grade 2: Anemia | 6 | 6
  Grade 2: Hemoglobin increased | 0 | 1
  Grade 2: Lymphocyte count decreased | 1 | 2
  Grade 2: Lymphocyte count increased | 6 | 9
  Grade 2: Neutrophil count decreased: number analyzed (Participants) | 209 | 204
  Grade 2: Neutrophil count decreased | 7 | 4
  Grade 2: White blood cell decreased | 1 | 0
  Grade 3: Anemia | 0 | 2

23. Secondary Outcome: Number of Participants With Chemistry Results by Maximum CTC Grade: TP2 and Beyond
Description: Blood samples were collected for analysis of clinical chemistry parameters: ALT increased, alkaline phosphatase increased (ALP), aspartate aminotransferase increased (AST), blood bilirubin increased, creatinine increased, hypercalcemia, hyperkalemia, hypernatremia, hypoalbuminemia, hypocalcemia, hypokalemia, hyponatremia. Laboratory parameters were graded according to NCI-CTC version 4.03 where, grade 0= within normal limits; Grade1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences and Grade 5: death. Categories with at least 1 non-zero value were reported.
Time Frame: Post randomization up to end of study treatment (maximum of 22 weeks)
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Switching Arm: Humira and PF-06410293 (Adalimumab) | Non-switching Arm: Humira (Adalimumab)
Number analyzed (Participants) | 212 | 208
Participants
  Grade 0: ALT increased: number analyzed (Participants) | 211 | 208
  Grade 0: ALT increased | 169 | 174
  Grade 0: ALP increased: number analyzed (Participants) | 211 | 208
  Grade 0: ALP increased | 202 | 196
  Grade 0: AST increased: number analyzed (Participants) | 211 | 208
  Grade 0: AST increased | 195 | 198
  Grade 0: Blood bilirubin increased: number analyzed (Participants) | 211 | 208
  Grade 0: Blood bilirubin increased | 205 | 204
  Grade 0: Creatinine increased: number analyzed (Participants) | 211 | 208
  Grade 0: Creatinine increased | 171 | 151
  Grade 0: Hypercalcemia: number analyzed (Participants) | 211 | 208
  Grade 0: Hypercalcemia | 211 | 207
  Grade 0: Hyperkalemia | 208 | 202
  Grade 0: Hypernatremia | 210 | 207
  Grade 0: Hypoalbuminemia | 212 | 208
  Grade 0: Hypocalcemia: number analyzed (Participants) | 211 | 208
  Grade 0: Hypocalcemia | 201 | 202
  Grade 0: Hypokalemia | 210 | 207
  Grade 0: Hyponatremia | 211 | 207
  Grade 1: ALT increased: number analyzed (Participants) | 211 | 208
  Grade 1: ALT increased | 40 | 33
  Grade 1: ALP increased: number analyzed (Participants) | 211 | 208
  Grade 1: ALP increased | 9 | 12
  Grade 1: AST increased: number analyzed (Participants) | 211 | 208
  Grade 1: AST increased | 16 | 10
  Grade 1: Blood bilirubin increased: number analyzed (Participants) | 211 | 208
  Grade 1: Blood bilirubin increased | 5 | 3
  Grade 1: Creatinine increased: number analyzed (Participants) | 211 | 208
  Grade 1: Creatinine increased | 39 | 52
  Grade 1: Hypercalcemia: number analyzed (Participants) | 211 | 208
  Grade 1: Hypercalcemia | 0 | 1
  Grade 1: Hyperkalemia | 4 | 6
  Grade 1: Hypernatremia | 2 | 1
  Grade 1: Hypocalcemia: number analyzed (Participants) | 211 | 208
  Grade 1: Hypocalcemia | 10 | 6
  Grade 1: Hyponatremia | 1 | 1
  Grade 2: ALT increased: number analyzed (Participants) | 211 | 208
  Grade 2: ALT increased | 2 | 1
  Grade 2: Blood bilirubin increased: number analyzed (Participants) | 211 | 208
  Grade 2: Blood bilirubin increased | 1 | 1
  Grade 2: Creatinine increased: number analyzed (Participants) | 211 | 208
  Grade 2: Creatinine increased | 1 | 5
  Grade 2: Hypokalemia | 2 | 1

24. Secondary Outcome: Number of Participants With Laboratory Results Based on Evaluation of Drug-Induced Serious Hepatotoxicity (eDISH) Analysis: TP2 and Beyond
Description: In this outcome measure, liver function laboratory parameters, which included: normal bilirubin and AST/ALT, Temple's Corollary (AST/ALT [more than or equal to] >=3*upper limit normal [ULN] and normal bilirubin), Gilbert's Syndrome or cholestasis (normal AST/ALT and bilirubin >=2*ULN) and Potential Hy's Law Cases (AST/ALT >=3*ULN and Bilirubin>=2*ULN) according to eDISH criteria, were reported.
Time Frame: Post randomization up to end of study treatment (maximum of 22 weeks)
Population: Safety randomized population included all participants who were randomized and received at least one dose of dose of investigational product following the randomization at Study Week 10. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Switching Arm: Humira and PF-06410293 (Adalimumab) | Non-switching Arm: Humira (Adalimumab)
Number analyzed (Participants) | 211 | 208
Participants
  Normal Bilirubin and AST/ALT | 208 | 207
  Temple's Corollary (AST/ALT >=3* upper limit normal [ULN] and Normal Bilirubin) | 2 | 1
  Gilbert's Syndrome or Cholestasis (Normal AST/ALT and Bilirubin >=2*ULN) | 1 | 0
  Potential Hy's Law Cases (AST/ALT >=3*ULN and Bilirubin>=2*ULN) | 0 | 0

25. Secondary Outcome: Baseline, Absolute Week 32 Values for Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP) and Change From Baseline in SBP, DBP at Week 32 (EOT/ ET)
Description: SBP and DBP were measured in a supine position using an automated device preceded by at least 5 minutes of rest for the participant in a quiet setting without any distractions. Baseline value was defined as the most recent measurement prior to the first dose of study treatment after randomization in TP2.
Time Frame: Baseline and Week 32 (end of treatment [EOT]/early termination [ET])
Population: Safety randomized population included all participants who were randomized and received at least one dose of study treatment following the randomization at Study Week 10. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Arm/Group | Switching Arm: Humira and PF-06410293 (Adalimumab) | Non-switching Arm: Humira (Adalimumab)
Number analyzed (Participants) | 212 | 209
Millimeter of mercury
  SBP: Baseline | 125.7 (12.72) | 125.9 (11.49)
  SBP: Absolute value at Week 32 (EOT/ET) | 126.0 (11.20) | 126.2 (12.69)
  SBP: Change at Week 32 (EOT/ET) | 0.3 (11.49) | 0.4 (11.28)
  DBP: Baseline | 78.1 (8.31) | 77.7 (7.60)
  DBP: Absolute value at Week 32 (EOT/ET) | 78.6 (7.77) | 77.5 (7.54)
  DBP: Change at Week 32 (EOT/ET) | 0.5 (8.04) | -0.2 (8.32)

26. Secondary Outcome: Baseline, Absolute Week 32 Values for Pulse Rate and Change From Baseline in Pulse Rate at Week 32 (EOT/ET)
Description: Pulse rate was measured in a supine position using an automated device preceded by at least 5 minutes of rest for the participant in a quiet setting without any distractions. Baseline value was defined as the most recent measurement prior to the first dose of study treatment after randomization in TP2.
Time Frame: Baseline and Week 32 (EOT/ET)
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Switching Arm: Humira and PF-06410293 (Adalimumab) | Non-switching Arm: Humira (Adalimumab)
Number analyzed (Participants) | 212 | 209
Beats per minute
  Baseline | 73.6 (8.55) | 73.2 (8.42)
  Absolute value at Week 32 (EOT/ET) | 73.6 (7.94) | 73.1 (7.98)
  Change at Week 32 (EOT/ET) | 0.1 (8.55) | -0.2 (7.68)

27. Secondary Outcome: Baseline, Absolute Week 32 Values for Temperature and Change From Baseline in Temperature at Week 32 (EOT/ET)
Description: Baseline value was defined as the most recent measurement prior to the first dose of study treatment after randomization in TP2.
Time Frame: Baseline and Week 32 (EOT/ET)
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Switching Arm: Humira and PF-06410293 (Adalimumab) | Non-switching Arm: Humira (Adalimumab)
Number analyzed (Participants) | 212 | 209
Degree Celsius
  Baseline | 36.5 (0.27) | 36.5 (0.27)
  Absolute value at Week 32 (EOT/ET) | 36.4 (0.26) | 36.4 (0.20)
  Change at Week 32 (EOT/ET) | -0.0 (0.28) | -0.0 (0.27)

28. Secondary Outcome: Baseline, Absolute Week 32 Values for Respiratory Rate and Change From Baseline in Respiratory Rate at Week 32 (EOT/ET)
Description: as for outcome 27
Time Frame: Baseline and Week 32 (EOT/ET)
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Switching Arm: Humira and PF-06410293 (Adalimumab) | Non-switching Arm: Humira (Adalimumab)
Number analyzed (Participants) | 212 | 209
Breaths per minute
  Baseline | 16.6 (1.75) | 16.6 (2.10)
  Absolute value at Week 32 (EOT/ET) | 16.5 (1.81) | 16.6 (2.00)
  Change at Week 32 (EOT/ET) | -0.1 (1.36) | -0.0 (1.52)

29. Secondary Outcome: Number of Participants Who Were Anti-Drug Antibodies (ADA) Positive and Neutralizing Antibodies (NAb) Positive
Description: Serum samples were analyzed using a validated electrochemoluminescent (ECL) immunoassay for ADA assessment. Samples positive for ADA were further tested for neutralizing activity using a validated cell based NAb assay. ADA positive was defined as ADA titer >=1.88 while NAb positive was defined as NAb titer >=0.70.
Time Frame: Week 10, 16, 22, 24, 26, 28, 32
Population: Safety randomized population included all participants who were randomized and received at least one dose of investigational product following the randomization at Study Week 10. For ADA: "Number Analyzed" = all participants assessed for ADA measurement at specific time points. For Nab: "Number Analyzed" = all participants with ADA positive results assessed for Nab measurement at specific time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Switching Arm: Humira and PF-06410293 (Adalimumab) | Non-switching Arm: Humira (Adalimumab)
Number analyzed (Participants) | 213 | 214
Participants
  Week 10: ADA positive | 55 | 59
  Week 10: NAb positive: number analyzed (Participants) | 55 | 59
  Week 10: NAb positive | 22 | 19
  Week 16: ADA positive | 88 | 97
  Week 16: NAb positive: number analyzed (Participants) | 88 | 97
  Week 16: NAb positive | 22 | 21
  Week 22: ADA positive | 96 | 106
  Week 22: NAb positive: number analyzed (Participants) | 96 | 106
  Week 22: NAb positive | 24 | 20
  Week 24: ADA positive | 102 | 100
  Week 24: NAb positive: number analyzed (Participants) | 102 | 100
  Week 24: NAb positive | 19 | 20
  Week 26: ADA positive | 101 | 105
  Week 26: NAb positive: number analyzed (Participants) | 101 | 105
  Week 26: NAb positive | 21 | 15
  Week 28: ADA positive | 102 | 105
  Week 28: NAb positive: number analyzed (Participants) | 102 | 105
  Week 28: NAb positive | 18 | 16
  Week 30: ADA positive | 103 | 109
  Week 30: NAb positive: number analyzed (Participants) | 103 | 109
  Week 30: NAb positive | 17 | 19
  Week 32: ADA positive | 100 | 104
  Week 32: NAb positive: number analyzed (Participants) | 100 | 104
  Week 32: NAb positive | 18 | 18

30. Secondary Outcome: Mean ADA Titers
Description: Serum samples were analyzed using a validated ECL immunoassay for ADA assessment. Endpoint titer was defined as log10 of the reciprocal of the ADA serum dilution at which the sample response was equal to the cut-point of the assay.
Time Frame: Week 10, 16, 22, 24, 26, 28, 30, 32
Population: Safety randomized population included all participants who were randomized and received at least one dose of investigational product following the randomization at Study Week 10. Here, 'Number Analyzed' signifies participants evaluable with ADA non-missing values at specific time points.
Measure: Mean (Standard Deviation); unit: log10 titer
Arm/Group | Switching Arm: Humira and PF-06410293 (Adalimumab) | Non-switching Arm: Humira (Adalimumab)
Number analyzed (Participants) | 213 | 214
log10 titer
  Week 10: number analyzed (Participants) | 211 | 214
  Week 10 | 0.830 (1.46534) | 0.880 (1.51789)
  Week 16: number analyzed (Participants) | 210 | 209
  Week 16 | 1.385 (1.71192) | 1.546 (1.75299)
  Week 22: number analyzed (Participants) | 208 | 202
  Week 22 | 1.570 (1.77364) | 1.784 (1.79136)
  Week 24: number analyzed (Participants) | 207 | 199
  Week 24 | 1.674 (1.78148) | 1.709 (1.78301)
  Week 26: number analyzed (Participants) | 204 | 198
  Week 26 | 1.671 (1.77780) | 1.806 (1.78134)
  Week 28: number analyzed (Participants) | 205 | 197
  Week 28 | 1.670 (1.77759) | 1.788 (1.77325)
  Week 30: number analyzed (Participants) | 206 | 198
  Week 30 | 1.658 (1.75135) | 1.854 (1.78187)
  Week 32: number analyzed (Participants) | 199 | 193
  Week 32 | 1.677 (1.76060) | 1.846 (1.81474)

31. Secondary Outcome: Mean NAb Titers
Description: Serum samples were analyzed using a validated ECL immunoassay for ADA assessment. Endpoint titer was defined as log10 of the reciprocal of the NAb serum dilution at which the sample response was equal to the cut-point of the assay.
Time Frame: Week 10, 16, 22, 24, 26, 28, 30, 32
Population: Safety randomized population included all participants who were randomized and received at least one dose of investigational product following the randomization at Study Week 10. Here, 'Number Analyzed' signifies participants evaluable with NAb non-missing values at specific time points.
Measure: Mean (Standard Deviation); unit: log10 titer
Arm/Group | Switching Arm: Humira and PF-06410293 (Adalimumab) | Non-switching Arm: Humira (Adalimumab)
Number analyzed (Participants) | 213 | 214
log10 titer
  Week 10: number analyzed (Participants) | 55 | 58
  Week 10 | 0.712 (1.02024) | 0.718 (1.14660)
  Week 16: number analyzed (Participants) | 88 | 97
  Week 16 | 0.467 (0.90051) | 0.443 (0.92450)
  Week 22: number analyzed (Participants) | 96 | 106
  Week 22 | 0.488 (0.91641) | 0.405 (0.89940)
  Week 24: number analyzed (Participants) | 102 | 100
  Week 24 | 0.396 (0.87759) | 0.409 (0.90030)
  Week 26: number analyzed (Participants) | 101 | 105
  Week 26 | 0.420 (0.90500) | 0.328 (0.84792)
  Week 28: number analyzed (Participants) | 102 | 105
  Week 28 | 0.360 (0.83177) | 0.353 (0.88464)
  Week 30: number analyzed (Participants) | 103 | 109
  Week 30 | 0.359 (0.87754) | 0.377 (0.91439)
  Week 32: number analyzed (Participants) | 100 | 104
  Week 32 | 0.341 (0.81482) | 0.362 (0.88055)

ADVERSE EVENTS:
Time Frame: TP1: Day 1 up to maximum of 10 Weeks TP2 and beyond: Post randomization up to maximum of 4 weeks after last dose (maximum of 26 weeks)
Description: Same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study. As planned, AE were analyzed for TP1 using the Safety-TP1 population for the Humira arm. AE analyses for TP2 and beyond were performed using Safety-randomized population for switching arm and non-switching arm.
Arm/Group | Humira (Adalimumab) | Switching Arm: Humira and PF-06410293 (Adalimumab) | Non-switching Arm: Humira (Adalimumab)
All-Cause Mortality (participants affected / at risk) | 0/445 | 0/213 | 0/214
Serious Adverse Events (participants affected / at risk) | 13/445 | 3/213 | 8/214
Other Adverse Events (participants affected / at risk) | 28/445 | 46/213 | 38/214
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Humira (Adalimumab) (N=445) | Switching Arm: Humira and PF-06410293 (Adalimumab) (N=213) | Non-switching Arm: Humira (Adalimumab) (N=214)
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 5 | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 1 | 1 | 2
Influenza (Infections and infestations) | 1 | 0 | 0
Lyme disease (Infections and infestations) | 2 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 | 0 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Keratitis (Eye disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Humira (Adalimumab) (N=445) | Switching Arm: Humira and PF-06410293 (Adalimumab) (N=213) | Non-switching Arm: Humira (Adalimumab) (N=214)
Injection site reaction (General disorders) | 13 | 6 | 4
Swelling (General disorders) | 0 | 3 | 1
Urinary tract infection (Infections and infestations) | 5 | 4 | 3
COVID-19 (Infections and infestations) | 0 | 16 | 9
Nasopharyngitis (Infections and infestations) | 0 | 0 | 7
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 3
SARS-CoV-2 test positive (Investigations) | 9 | 18 | 14
Alanine aminotransferase increased (Investigations) | 0 | 3 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 3 | 1
Erythema (Skin and subcutaneous tissue disorders) | 10 | 6 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
Headache (Nervous system disorders) | 0 | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Hypertension (Vascular disorders) | 0 | 2 | 5

LIMITATIONS AND CAVEATS:
In participant flow, there were discontinuations due to AEs, which were captured within different reasons for discontinuations (e.g. other, physician decision etc.) as the study case report form (CRF) page did not include AE as an option for sites to record if the discontinuation was truly due to AE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from the study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/13/NCT04230213/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-13): https://cdn.clinicaltrials.gov/large-docs/13/NCT04230213/SAP_001.pdf